CLINICAL TRIAL: NCT03121976
Title: Comparison of Continuous Femoral Nerve Block Using Ultrasound Versus Ultrasound and Nerve Stimulation Using Stimulating Catheter in Patients Undergoing Total Knee Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: A Comparison of US and Evoked Motor Response-guided Placement of Continuous Femoral Nerve Block Following TKA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 373-2011
Record Dates: First submitted 2017-04-04; First posted 2017-04-20 (Actual); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Anesthesia; Pain; Nerve Pain; Knee Arthroplasty; Nerve Block
MeSH Terms: conditions — Pain; Neuralgia | interventions — Ultrasonography

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound (Experimental): Femoral catheters inserted using ultrasound only
  Interventions: Device: Ultrasound
- Ultrasound + Nerve Stimulation (Active Comparator): Femoral catheters inserted using ultrasound with nerve stimulation
  Interventions: Device: Ultrasound + Nerve Stimulation

INTERVENTIONS:
Device: Ultrasound — Femoral catheter inserted using ultrasound only
  Arms: Ultrasound
Device: Ultrasound + Nerve Stimulation — Femoral catheter inserted using ultrasound and nerve stimulation
  Arms: Ultrasound + Nerve Stimulation

SUMMARY:
The purpose of this study is to determine which technique for catheter placement in continuous femoral nerve block (FNB) is most successful - guidance with (1) ultrasound or (2) nerve stimulation and ultrasound. Sensory and motor assessment scores will be obtained post-FNB. Patient controlled analgesia and opiate consumption is also recorded along with pain scores for the first 48 hour post-FNB.

DETAILED DESCRIPTION:
Continuous femoral nerve block (cFNB) is a widely used regional anesthetic technique for many lower limb operations, such as total knee arthroplasty (TKA), anterior cruciate ligament repair, tibial osteotomy and patellar surgery. It provides superior pain relief, faster ambulation, shorter hospital stays and less risk of side effects in comparison to patient controlled analgesia (PCA), local anesthetic wound infiltration, or single shot femoral nerve block (FNB).

Stimulating catheters were introduced in 1999 to provide an objective end point to guide continuous nerve block catheter position by maintaining the desired evoked muscle response with nerve stimulation (NS). The main advantages of stimulating catheters are faster onset of sensory and motor block and reduction of local anesthetic drugs consumption. In recent years the precise insertion of continuous catheters has improved especially with the introduction of ultrasound (US)-guided imaging to regional anesthesia practice and advances in scanning techniques. That led to a call to reduce cost by switching to non-stimulating catheters. However, most studies comparing both catheters lacked anesthetic technique standardization and adequate sample size.

In this prospective randomized controlled trial, we compared postoperative analgesic efficacy and opioids consumption in patients having cFNB insertion using US alone and that of US combined with NS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status I to III patients
* Aged 18-75 scheduled for unilateral TKA

Exclusion Criteria:

* History of significant psychiatric problems
* BMI > 40 kg/m^2
* Prior surgery in the inguinal region
* Neurological disease with sensory or motor deficit
* Diabetic neuropathy
* Contraindication to any study medications
* Daily opioid consumption >10 mg PO morphine (or equivalent) for 2 weeks prior to surgery

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2012-01-02 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2013-03-31 (Actual)

PRIMARY OUTCOMES:
Mean numeric pain score (NRS) | 24 hours post-block insertion
  Pain score assessed 24 hours post-block insertion using numeric pain scale from 0-10

SECONDARY OUTCOMES:
Time to perform the block | At the time of block procedure
  Time required to perform the block procedure
Sensation over the skin of the thigh to determine sensory block using 3 point grading scale | 30 min post-block insertion
  Sensory block evaluation examined the sensation over the skin of the thigh
Quadriceps muscle strength to determine motor block using 3 point grading scale | 30 min post-block insertion
  Motor block evaluation examined quadriceps muscle strength by grading the ability or inability to extend the leg of the limb to be operated on against gravity after the hip is passively flexed at 45°
Total hydromorphone used (oral and intravenous PCA) | 24 hours post-block
  Total amount of hydromorphone consumed within 24 hours post-block
Total hydromorphone used (oral and intravenous PCA) | 48 hours post-block
  Total amount of hydromorphone consumed within 48 hours post-block

CONTACTS AND LOCATIONS:
Overall Officials: Imad Awad, MBChB, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pham Dang C, Lelong A, Guilley J, Nguyen JM, Volteau C, Venet G, Perrier C, Lejus C, Blanloeil Y. Effect on neurostimulation of injectates used for perineural space expansion before placement of a stimulating catheter: normal saline versus dextrose 5% in water. Reg Anesth Pain Med. 2009 Sep-Oct;34(5):398-403. doi: 10.1097/AAP.0b013e3181b48648. PMID 19920414
- [Background] Dauri M, Fabbi E, Mariani P, Faria S, Carpenedo R, Sidiropoulou T, Coniglione F, Silvi MB, Sabato AF. Continuous femoral nerve block provides superior analgesia compared with continuous intra-articular and wound infusion after anterior cruciate ligament reconstruction. Reg Anesth Pain Med. 2009 Mar-Apr;34(2):95-9. doi: 10.1097/AAP.0b013e31819baf98. PMID 19282706
- [Background] Paul JE, Arya A, Hurlburt L, Cheng J, Thabane L, Tidy A, Murthy Y. Femoral nerve block improves analgesia outcomes after total knee arthroplasty: a meta-analysis of randomized controlled trials. Anesthesiology. 2010 Nov;113(5):1144-62. doi: 10.1097/ALN.0b013e3181f4b18. PMID 20966667
- [Background] Shum CF, Lo NN, Yeo SJ, Yang KY, Chong HC, Yeo SN. Continuous femoral nerve block in total knee arthroplasty: immediate and two-year outcomes. J Arthroplasty. 2009 Feb;24(2):204-9. doi: 10.1016/j.arth.2007.09.014. Epub 2008 Mar 4. PMID 18534496
- [Background] Carli F, Clemente A, Asenjo JF, Kim DJ, Mistraletti G, Gomarasca M, Morabito A, Tanzer M. Analgesia and functional outcome after total knee arthroplasty: periarticular infiltration vs continuous femoral nerve block. Br J Anaesth. 2010 Aug;105(2):185-95. doi: 10.1093/bja/aeq112. Epub 2010 Jun 14. PMID 20551021
- [Background] Salinas FV, Liu SS, Mulroy MF. The effect of single-injection femoral nerve block versus continuous femoral nerve block after total knee arthroplasty on hospital length of stay and long-term functional recovery within an established clinical pathway. Anesth Analg. 2006 Apr;102(4):1234-9. doi: 10.1213/01.ane.0000198675.20279.81. PMID 16551930
- [Background] Boezaart AP, de Beer JF, du Toit C, van Rooyen K. A new technique of continuous interscalene nerve block. Can J Anaesth. 1999 Mar;46(3):275-81. doi: 10.1007/BF03012610. PMID 10210055
- [Background] Martinez Navas A, Vazquez Gutierrez T, Echevarria Moreno M. Continuous lateral popliteal block with stimulating catheters. Acta Anaesthesiol Scand. 2005 Feb;49(2):261-3. doi: 10.1111/j.1399-6576.2004.00574.x. PMID 15715632
- [Background] Casati A, Fanelli G, Koscielniak-Nielsen Z, Cappelleri G, Aldegheri G, Danelli G, Fuzier R, Singelyn F. Using stimulating catheters for continuous sciatic nerve block shortens onset time of surgical block and minimizes postoperative consumption of pain medication after halux valgus repair as compared with conventional nonstimulating catheters. Anesth Analg. 2005 Oct;101(4):1192-1197. doi: 10.1213/01.ane.0000167232.10305.cd. PMID 16192543
- [Background] Cappelleri G, Ghisi D, Ceravola E, Guzzetti L, Ambrosoli AL, Gemma M, Cornaggia G. A randomised controlled comparison between stimulating and standard catheters for lumbar plexus block. Anaesthesia. 2015 Aug;70(8):948-55. doi: 10.1111/anae.13077. Epub 2015 Mar 21. PMID 25810108